CLINICAL TRIAL: NCT03940898
Title: A Follow-up Study of Clinical Effects of Repetitive Transcranial Magnetic Stimulation on Schizophrenia
Brief Title: The Mid-term Effect of Repeated Transcranial Magnetic Stimulation on Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JCai
Record Dates: First submitted 2019-04-29; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Schizophrenia
Keywords: Repetitive transcranial magnetic stimulation; Schizophrenia; Cerebellar vermis; Negative symptoms; Depressive symptoms; Cognitive function; Follow-up study
MeSH Terms: conditions — Schizophrenia; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group-active rTMS (Active Comparator): Participants in the study group received 100%MT(motor threshold) repetitive transcranial magnetic stimulation with the intermittent theta burst stimulation paradigm.
  Interventions: Device: repetitive transcranial magnetic stimulation
- control group-shame rTMS (Sham Comparator): Participants in the control group received rTMS pseudo-stimulation intervention. The stimulation head was inverted by 180 degrees or 90 degrees according to the model of the stimulation device to achieve pseudo-stimulation and the remaining stimulation parameters were consistent with the study group.
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — There are two types of stimulation equipment, one is the transcranial magnetic stimulator model Magpro X100 produced by Danish Medtronic, and the other is the CCY-I TMS stimulator produced by Wuhan Eride, model B9076. The stimulating magnetic head uses an "8" shaped coil, and the stimulation site is the cerebellar vermis (ie, 1 cm below the occipital bulge), and the stimulation intensity is 100% of the motor threshold.The base frequency of the iTBS mode is 5 Hz, and one short burst stimulus occurs every 200 milliseconds. In each short array, three single pulses with a frequency of 50 Hz are buried, and each 10 short burst stimulation intervals are 8 seconds, for a total of 200 short burst stimulations. The total number of stimulation pulses is 600 per day.It takes 3 minutes and 20 seconds to complete one intervention. All participants were intervened once a day for 5 times a week for 2 weeks for a total of 10 times.

SUMMARY:
Medications have a poor effect on negative symptoms and cognitive function in schizophrenia. In the past, most of the studies on repetitive transcranial magnetic stimulation intervention in patients with schizophrenia used conventional stimulation sites and patterns, and the intervention effect was still controversial. A few studies have achieved positive results with the new stimulation model (TBS model) and the therapeutic target (cerebellar vermis), but the follow-up period did not exceed 2 weeks, and no similar studies have emerged in China. Therefore, this study hypothesized that the TBS-mode rTMS intervention in the cerebellar vermis can improve the negative symptoms, cognitive function, and depressive symptoms of schizophrenia, and the efficacy can be maintained.

DETAILED DESCRIPTION:
Medications have a poor effect on negative symptoms and cognitive function in schizophrenia. In the past, most of the studies on repetitive transcranial magnetic stimulation intervention in patients with schizophrenia used conventional stimulation sites and patterns, and the intervention effect was still controversial. A few studies have achieved positive results with the new stimulation model (TBS model) and the therapeutic target (cerebellar vermis), but the follow-up period did not exceed 2 weeks, and no similar studies have emerged in China. Therefore, this study hypothesized that the TBS-mode rTMS intervention in the cerebellar vermis can improve the negative symptoms, cognitive function, and depressive symptoms of schizophrenia, and the efficacy can be maintained.

1. Aim of the study: 1.1 To explore the clinical efficacy of cerebellar vermal theta burst stimulation for negative symptoms, cognitive function and depressive symptoms in patients with schizophrenia. 1.2 The patients were followed up for 24 weeks to explore the duration of rTMS efficacy
2. Introduction of the study: This is a multi-center, randomized, sham-controlled, double-blinded trial. Participants diagnosed with schizophrenia from Shanghai Mental Health Center and six district-level mental health centers were randomized according to the odd-even sequence of enrollment, with odd numbers into the study group and even numbers into the control group. Patients in the study group received 100%MT rTMS with the intermittent theta burst stimulation paradigm, while another patients were subjected to pseudo-stimulation treatment, both being given 2-week intervention (5 times per week). The type and dose of antipsychotic drugs taken by patients remained unchanged during the intervention period. Efficacy were assessed with the Positive and Negative Symptoms Scale (PANSS), Hamilton Depression Scale (HAMD-24) and MATRICS Consensus Cognitive Battery (MCCB).

ELIGIBILITY:
Inclusion Criteria:

* the patient met the diagnostic criteria for schizophrenia in ICD-10;
* 18-50 years old;
* Right handed;
* The current condition is stable, and the types and doses of antipsychotic drugs are unchanged;
* In the PANSS scale, the score of Pl, P3, P5, P6, and G9 is not more than 5 points, and the score of P2 is not more than 4 points;

Exclusion Criteria:

* In addition to schizophrenia, patients with other mental illnesses；
* Contraindications to rTMS;
* Patients receiving ECT(electro-convulsive therapy) in last month;
* Pregnant or lactating woman.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
PANSS-N | 24 weeks
  The efficacy of negative symptoms was assessed based on the patient's score changes on the PANSS（Positive and Negative Syndrome Scale） negative symptom subscale. PANSS is a relatively mature assessment tool commonly used in clinical research to assess the severity of schizophrenia symptoms. It consists of a positive symptom subscale (7 items), a negative symptom subscale (7 items) and a general psychopathological symptom subscale (16 items), a total of 30 items.Each item has specific definitions and operational grading criteria. It is divided into 7 grades according to the level of psychopathology (1~7 points). The higher the score, the heavier the symptoms. The total score of PANSS is 30- 210 points, the positive symptom subscale and the negative symptom subscale are 7-49 points, and the general psychopathological symptoms subscale is 16 to 112 points.

SECONDARY OUTCOMES:
MCCB | 24 weeks
  The efficacy of cognitive function was assessed based on the patient's score changes on MCCB（MATRICS Consensus Cognitive Battery）.MCCB is a set of neuropsychological tests specifically designed to assess cognitive function in schizophrenia. The MCCB Chinese version includes 9 subtests: Train Making Test, Brief Assessment of Cognition in Schizophrenia, Hopkins Verbal Learning Test, Wechsler Working Memory, Neuropsychological Assessment Battery: Mazes, Brief visuospatial Memory Test, Categoary Fluency (Animal Naming), MSCEIT Emotional Intelligence Test, Continuous Performance Test-Identical Pairs. After the test, the MCCB computer scoring program is used to convert the rough points of each subtest into T scores, and the overall comprehensive score is calculated by the software. The range of each test and the overall composite score T is 0-100 points. The lower the score, the worse the cognitive function.
HAMD-24 | 24 weeks
  The efficacy of depressive symptoms was assessed based on the patient's total score changes on HAMD(Hamilton Depression Scale).This study used the 24 version of HAMD. Most of the items in the scale use a five-level scoring standard. The score of each item is between 0 and 4 points, with 0 points representing no; 1 point being mild; 2 points being moderate; 3 points being severe; 4 points being extremely severe. A small number of items use a three-level scoring standard, the score of each item is between 0 and 2 points, with 0 points representing no; 1 point being light-moderate; 2 points being severe. The higher the score, the more severe the symptoms. The total score of the scale ranges from 0 to 76 points.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cai, Study Director — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No